CLINICAL TRIAL: NCT01018914
Title: A Randomized, Open-Label, Comparative, Multi-Center Study to Assess the Safety and Efficacy of Prograf® (Tacrolimus)/ Myfortic® and Advagraf® (Extended Release Tacrolimus) / Myfortic® in de Novo Liver Transplant Recipients
Brief Title: A Study to Compare Safety and Efficacy of Prograf + Myfortic and Advagraf + Myfortic in Liver Transplantation Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVLTx-0901-TW
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Liver Transplantation
Keywords: Prograf; Advagraf; Myfortic
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf with Myfortic (Active Comparator)
  Interventions: Drug: Prograf; Drug: Myfortic
- Advagraf with Myfortic (Experimental)
  Interventions: Drug: Advagraf; Drug: Myfortic

INTERVENTIONS:
Drug: Prograf — oral
  Other Names: Tacrolimus; FK506
  Arms: Prograf with Myfortic
Drug: Advagraf — oral
  Other Names: Extended release tacrolimus; FK506E; MR4
  Arms: Advagraf with Myfortic
Drug: Myfortic — oral
  Other Names: Mycophenolate sodium

SUMMARY:
To compare the safety and efficacy of Prograf® with Myfortic® to Advagraf® extended release tacrolimus with Myfortic® in de novo liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a primary liver transplant recipient
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to transplant
* Patient has been fully informed and has signed an IRB approved informed consent form and is willing and able to follow study procedures
* Patient must receive 1st dose of study drug within 24 hours of pre-transplantation

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a liver
* Patient currently requires dialysis
* Patient has received a liver transplant from a non-heart beating donor
* Patient has received an ABO incompatible donor liver
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Patient has fulminant hepatic failure, unless hemodynamically stable
* Patient has an uncontrolled concomitant infection, a systemic infection requiring treatment (except viral hepatitis), or any other unstable medical condition that could interfere with the study objectives
* Patient is currently taking or has been taking an investigational drug in the 30 days prior to transplant
* Patient has a known hypersensitivity to tacrolimus, enteric-coated mycophenolate sodium or corticosteroids
* Patient is pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy confirmed acute rejection | during the 6 months post-transplant.

SECONDARY OUTCOMES:
Patient and graft survival rates | during the 6 months post-transplant
Time to first biopsy confirmed acute rejection episode | during the 6 months post-transplant
Incidence of anti-lymphocyte antibody therapy for treatment of rejection | during the 6 months post-transplant.
Safety assessed by adverse events, laboratory parameters, physical examinations and vital signs | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (3):
- Taiwan (3):
  - Taichung
  - Tainan
  - Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=ADVLTx-0901-TW